CLINICAL TRIAL: NCT02670590
Title: NAFLD: Independent Effects of Western Dietary Pattern Profile and Sedentary Life
Acronym: ct-NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Guglielmo Trovato, MD, PhD, Dirigente Medico, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOVE
Record Dates: First submitted 2016-01-15; First posted 2016-02-02 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NAFLD (Experimental): diet
  Interventions: Behavioral: diet

INTERVENTIONS:
Behavioral: diet — diet

SUMMARY:
Investigators perform a counseling intervention study (6 months) in adult subjects with evidence of Fatty Liver by Ultrasound, graded 0-3 according to the Bright Liver Score (BLS); exclusion criteria are diabetes, renal insufficiency (glomerular filtration rate < 90 ml/min), cancer, heart failure > II NYHA ( New York Heart Association) Class), chronic virus hepatitis, and cirrhosis. Insulin resistance was assessed as homeostasis model assessment-insulin resistance (HOMA-IR) . Suggestions and advice on individual "healthy" food purchase, storage, and cooking were given. Reliable feedback and evidence of patients' adherence were obtained by scheduled dietician's interviews. Investigators will challenge the predictive effects of the Adherence to Mediterranean Diet, of Western dietary profile score and of increased physical activity at 6 months in a body mass index changes-balanced model to detect independent effects, if any, of the studied variable on NAFLD persistence, amelioration or disappearance. Threshold and odds of Mediterranean and Western dietary profile score will be calculated by contingency tables and receiver operator characteristic curve (ROC) analysis..

DETAILED DESCRIPTION:
Dietary and physical exercise counseling.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of fatty liver

Exclusion Criteria:

* type I or type II diabetes,
* no alcohol, cancer, malnutrition, severe obesity, renal insufficiency, viral hepatitis, other chronic disease

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Decrease of fatty liver appearance by ultrasound | 6 months

IPD SHARING:
Plan to Share IPD: Undecided